CLINICAL TRIAL: NCT05207722
Title: A Phase I/IIa Open Label, Non-Randomized, Multicenter Study of CYNK-101 in Combination with Trastuzumab and Pembrolizumab in Patients with Locally Advanced Unresectable or Metastatic HER2-Positive Gastric or Gastroesophageal Junction (G/GEJ) Aenocarcinoma
Brief Title: CYNK-101 in Combination with Trastuzumab and Pembrolizumab in Patients with Locally Advanced Unresectable or Metastatic HER2-Positive Gastric or Gastroesophageal Junction (G/GEJ) Adenocarcinoma
Status: Terminated | Phase: Phase 1 / Phase 2 | Type: Interventional
Why Stopped: for business reasons
Sponsor: Celularity Incorporated (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Sequential | Masking: None | Purpose: Treatment
Other Study IDs: CYNK-101-HER2-001
Record Dates: First submitted 2022-01-12; First posted 2022-01-26 (Actual); Last update posted 2024-12-12 (Actual); Status verified 2024-02

CONDITIONS: Metastatic HER2 Positive Gastroesophageal Junction Cancer
Keywords: CYNK-101; Natural Killer Cells; Cell Therapy; Metastatic HER2-positive Gastric Cancer; Gastric Cancer; Gastroesophageal Junction Adenocarcinoma
MeSH Terms: conditions — Stomach Neoplasms | interventions — pembrolizumab; Trastuzumab; aldesleukin; Cyclophosphamide; fludarabine; fludarabine phosphate; Mesna

STUDY DESIGN:
Intervention Model Description: This Phase I/IIa study will utilize a 3+3 open label design, and will evaluate two escalating dosing Cohort levels of CYNK-101 in combination with rhIL2 following and initial induction and lymphodepletion regimen. Once the Maximum Tolerated Dose (MTD) or Recommended Phase 2 Dose (RP2D) is determined in Phase I, the Phase IIa portion of the study will commence.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (2):
- Phase I Dose Escalation (Experimental): Up to two dosing cohorts of CYNK-101 in combination with rhIL2 will be evaluated following an initial induction and lymphodepletion regimen.
  Interventions: Biological: CYNK-101; Drug: Pembrolizumab; Drug: Trastuzumab; Drug: Recombinant Human Interleukin-2; Drug: Cyclophosphamide; Drug: Fludarabine; Drug: Mesna
- Phase IIa Expansion (Experimental): Once the Maximum Tolerated Dose (MTD) or Recommended Phase 2 Dose (RP2D) is determined in Phase I, the Phase IIa portion of the study will commence.
  Interventions: Biological: CYNK-101; Drug: Pembrolizumab; Drug: Trastuzumab; Drug: Recombinant Human Interleukin-2; Drug: Cyclophosphamide; Drug: Fludarabine; Drug: Mesna

INTERVENTIONS:
Biological: CYNK-101 — CYNK-101 is a human placental hematopoietic stem/progenitor cell derived NK cell product, that is genetically modified to express a variant of CD16, Fc gamma receptor III (FcγRIII).
Drug: Pembrolizumab — 200 mg on Day 1 of each 3-week cycle as an IV infusion.
  Other Names: Keytruda®
Drug: Trastuzumab — 8 mg/kg loading dose and then 6 mg/kg maintenance dose administered IV on day 1 of each 3-week cycle.
  Other Names: Herceptin®
Drug: Recombinant Human Interleukin-2 — 6 million (M) international units (IU) of rhIL-2 administered subcutaneously (SC) on each CYNK-101 infusion day.
  Other Names: proleukin
Drug: Cyclophosphamide — Cyclophosphamide: 900 mg/m2 administered IV as part of a 3-day lymphodepletion regimen.
  Other Names: cytoxan
Drug: Fludarabine — Fludarabine: 30 mg/m2 administered IV as part of a 3-day lymphodepletion regimen.
  Other Names: fludara
Drug: Mesna — MESNA: shall be administered as part of a 3-day lymphodepletion regimen for the inhibition of hemorrhagic cystitis induced by cyclophosphamide. Route of administration, dosage, and frequency of Mesna should be based on institutional standards.

SUMMARY:
This study will find the maximum tolerated dose (MTD) of CYNK-101 which contains Natural Killer (NK) cells derived from human placental CD34+ cells and culture-expanded. CYNK-101 will be administered as first-line treatment, following induction therapy consisting of Pembrolizumab, Trastuzumab and a Fluoropyrimidine / Platinum based Chemotherapy regimen. Patients are required to undergo a biopsy for confirmation of HER2 positivity defined as either IHC 3+ or IHC 2+ with a positive fluorescent in-situ hybridization (FISH) or FISH + alone. The safety of this treatment will be evaluated, and researchers will want to learn if NK cells will help in treating patients with Locally Advanced Unresectable or Metastatic HER2-Positive Gastric or Gastroesophageal Junction (G/GEJ) Adenocarcinoma.

ELIGIBILITY:
Inclusion Criteria:

1. Be at least 18 years of age on the day of signing informed consent.
2. Have cytologically or histologically confirmed diagnosis for the first-line treatment of patients with locally advanced unresectable or metastatic HER2-Positive Gastric or Gastroesophageal junction (G/GEJ) adenocarcinoma.

   • Patients who have received adjuvant therapy more than 12 months prior to Visit 2 will be allowed to participate in the study. Any patient who has completed an INDUCTION regimen prior to study entry and achieved best tumor response as either (1) Stable Disease per RECIST after 6 cycles or (2) Progressive Disease per RECIST and meets all other inclusion/exclusion criteria per protocol, will be eligible for enrollment in this clinical trial to continue with LYMPHODEPLETION and NK CELL INDUCTION and MAINTENANCE.
3. Patients will be required to undergo a biopsy for confirmation of HER2 expression prior to study entry.

   * HER2 overexpression is defined by immunohistochemistry (IHC) or in situ hybridization (ISH) for amplification of HER2 gene.
   * Patients must have either IHC 3+ or IHC 2+ with a positive fluorescent in-situ hybridization (FISH) or FISH + alone, as assessed locally on primary or metastatic tumor.
   * Due to differences in tumor histopathology, use of FDA-approved tests, specific for Gastric Cancers, will be required when assessing HER2 Expression [HERCEPTIN package insert; 202120].
4. Have measurable disease as assessed by the investigator according to RECIST 1.1 [Eisenhauer EA et al, 200913].
5. Have a performance status of 0-1 on the Eastern Cooperative Oncology Group (ECOG) performance scale.
6. Have a life expectancy of ≥ 6 months.
7. Patients must agree to use a highly effective method of contraception from the start of the study until 1 year after the last dose of lymphodepletion or 4 months from last dose of pembrolizumab, or 6 months from last dose of trastuzumab; whichever comes later.
8. Have adequate cardiac function, defined as left ventricular ejection fraction > 45% as determined by MUGA scan or ECHO and QT interval calculated according to the Fridericia method (≤ 470 ms for men and ≤480 ms for women).
9. Demonstrate adequate organ function by laboratory values as follows:

   * Hematological:

     * Absolute neutrophil count (ANC) ≥ 1.5 x 109/L,
     * Platelet count ≥ 100 x 109/L
     * Hemoglobin ≥ 9 g/dL or ≥ 5.6 mmol/L
   * Renal:

     o Calculated creatinine clearance (Cockcroft-Gault Formula) ≥ 50 mL/min
   * Hepatic:

     o Total bilirubin ≤1.5 x ULN
     * Exception: Patients with Gilbert's disease total bilirubin ≤ 3.0 x ULN

       o Aspartate aminotransferase (AST) and alanine aminotransferase (ALT) ≤ 2.5 x ULN
     * Exception: AST and ALT ≤ 5 x ULN for patients with liver metastases.
   * Coagulation:

     * Prothrombin Time (PT) ≤ 1.5 x ULN unless patient is receiving anticoagulant therapy if PT or PTT is within therapeutic range of intended use of anticoagulants
     * activated Partial Thromboplastin Time (aPTT) ≤ 1.5 x ULN unless patient is receiving anticoagulant therapy if PT or PTT is within therapeutic range of intended use of anticoagulants

Exclusion Criteria:

1. Patients who have received prior systemic therapy for locally advanced unresectable or metastatic disease.
2. Has had major surgery, open biopsy, or significant traumatic injury within 28 days prior to Visit 2, or anticipation of the need for major surgery during the course of study treatment.
3. Has had radiotherapy within 14 days prior to Visit 2.
4. Has a known additional malignancy that is progressing or has required active treatment within the past 3 years.

   • Exceptions: Squamous or Basal cell carcinoma of the skin, superficial bladder cancer, and prostate cancer not requiring treatment.
5. Patients with symptomatic, untreated, or actively progressing CNS metastases. Patients with a history of CNS metastases are eligible if they have not received radiotherapy within 7 days or whole-brain radiation for the past 14 days. Patients should not be receiving ongoing treatment with either corticosteroids or anticonvulsants. Patients with new CNS metastases detected during the Screening period, may participate in the study if they receive radiotherapy or surgery resulting in stable metastatic disease.
6. Has an active autoimmune disease that has required systemic treatment in the past 2 years.
7. Patients with hypothyroidism who are on stable replacement therapy will be allowed.
8. Has a diagnosis of immunodeficiency or is receiving chronic systemic steroid therapy greater than 10 mg per day of prednisone or equivalent.

   • Patients who require replacement for adrenal insufficiency will be allowed.
9. Has a history of (non-infectious) pneumonitis that requires steroids or current pneumonitis.
10. Has a known history of active tuberculosis.
11. Has an active infection requiring systemic therapy.
12. Accumulation of pleural, ascitic, or pericardial fluid requiring drainage or diuretic drugs within 14 days prior to Visit 2. If the participant is receiving diuretic drugs for other reasons, it is acceptable.
13. Has peripheral neuropathy > Grade 1.
14. Has a known psychiatric or substance abuse disorder that would interfere with cooperation with the requirements of the trial.
15. Has active or clinically significant cardiac disease including:

    * History of myocarditis
    * History or presence of serious uncontrolled cardiac arrhythmias.
    * Clinically significant resting bradycardia.
    * Left ventricular ejection fraction (LVEF) as determined by echocardiogram (ECHO) < 45% or multiple gated acquisition scan (MUGA) < 45%.
    * Any of the following within 6 months prior to the start of the study treatments:

    myocardial infarction (MI), severe/unstable angina, congestive heart failure (CHF), cerebrovascular accident (CVA), transient ischemic attack (TIA).
16. Patients with history of human immunodeficiency virus (HIV) infection must be seronegative.
17. Known active infection with hepatitis B, hepatitis C, SARS-CoV-2, or other viral infections requiring systemic therapy.
18. Patients having a potential hypersensitivity (≥ Grade 3) to pembrolizumab, trastuzumab, study chemotherapy agents, rhIL-2 and/or to any excipients, murine proteins, or platinum-containing products. NOTE: any adverse events which has occurred because of prior therapy MUST have resolved to ≤ Grade 1 according to CTCAE (NCI Common Terminology Criteria for Adverse Events) Version 5 prior to study entry.
19. Has had an allogeneic tissue/solid organ transplant.
20. Immunized with live vaccine ≤ 28 days before Visit 2.
21. Participation in study of investigational agent or device ≤ 28 day prior to Visit 2.
22. Patient is pregnant or breastfeeding.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 1 (Actual)
Dates: Start 2022-04-14 (Actual); Primary Completion 2024-02-15 (Actual); Study Completion 2024-02-15 (Actual)

PRIMARY OUTCOMES:
Dose-Limiting Toxicity (DLT) | up to 28 days
  Phase I
Maximum Tolerated Dose (MTD) | up to 28 days
  Phase I
Overall Response Rate (ORR) as determined by the RECIST 1.1 Investigator using RECIST 1.1. | up to 12 months
  Phase IIa

SECONDARY OUTCOMES:
Progression Free Survival (PFS) | at 6 and 12 months
  Phase I/IIa
Duration of Response (DoR) | up to 12 months
  Phase I/IIa
Overall Response Rate (ORR) as determined by the RECIST 1.1 | up to 12 months
  Phase I
Incidence of Response conversion post CYNK-101 infusion | up to 12 months
  Phase I/IIa
Incidence of Treatment Emergent adverse events (TEAE) | up to 12 months
  Phase I/IIa
Incidence and Severity of adverse events (AEs) and clinically significant changes in laboratory values | up to 12 months
  Phase I/IIa
Incidence of replication competent lentivirus (RCL) | up to 12 months
  Phase I/IIa
Overall Survival (OS) | up to 12 months
  Phase I/IIa

CONTACTS AND LOCATIONS:
Overall Officials: Adrian Kilcoyne, MD, Study Director — Celularity Incorporated
Locations (3):
- United States (3):
  - Scripps Health, La Jolla, California
  - Georgetown, Washington D.C., District of Columbia
  - John Theurer Cancer Center at Hackensack University Medical Center, Hackensack, New Jersey

IPD SHARING:
Plan to Share IPD: No